CLINICAL TRIAL: NCT03501810
Title: Prospective, Single-Arm, Post-Market Clinical Follow-up (PMCF) Study to Further Assess the Safety and Performance of the OrtoWell® Distractor in Patients Undergoing Spinal Surgery
Brief Title: Study Assessing Safety and Performance of OrtoWell Distractor in Patients Undergoing Spinal Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: OrtoWay AB (Industry)
Collaborators: MedPass International (Industry)
Responsible Party: Sponsor
Other Study IDs: 01-2017
Record Dates: First submitted 2018-03-12; First posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Spinal Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Distractor use for vertebrae separation — Distractor use where separation of vertebrae is required, including corpectomy, insertion of disc prosthesis, insertion of an anterior lumbar interbody fusion (ALIF) cage, and tumor surgery

SUMMARY:
Study to Assess the Safety and Performance of the OrtoWell® Distractor in Patients Undergoing Spinal Surgery

DETAILED DESCRIPTION:
This is a Prospective, single-arm, multi-center, observational, post-market clinical follow-up study The OrtoWell® Distractor System (CE marked) is a device intended for separating and holding apart vertebral bodies in the spinal column, to facilitate removal of damaged discs, and implantation of disc prostheses or spinal cage prostheses, as well as for repositioning the vertebral bodies following implantation of disc or cage prostheses The OrtoWell® Distractor System will be used in patients undergoing anterior or lateral spinal surgery, where separation of vertebrae is required, including corpectomy, insertion of disc prosthesis, insertion of an anterior lumbar interbody fusion (ALIF) cage, and tumor surgery The study will enroll up to 32 patients in Germany that require one of the above listed intervention except the patients with a known osteoporosis Study subjects are expected to participate for approximately 30 days following the surgery. Participation will involve a screening period, surgery and scheduled follow-up assessment at 30 days post implant

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing spinal surgery, where use of the OrtoWell® Distractor System is indicated
* Signed written informed consent

Exclusion Criteria:

* Pregnant patients at the time of spinal surgery
* Known osteoporosis
* BMI ≥ 30
* Obstacles to performing radioscopy (primarily lateral), such as obesity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing anterior or lateral spinal surgery, where separation of vertebrae is required, including corpectomy, insertion of disc prosthesis, insertion of an anterior lumbar interbody fusion (ALIF) cage, and tumor surgery
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2018-04-05 (Actual); Primary Completion 2018-07-31 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Device Reliability | During the procedure
  Assessed by positioning accuracy,holding capability and ease of use

SECONDARY OUTCOMES:
Length of Procedure (hours) | During the procedure
  Length of Procedure
Major complications | Intra and peri operative periods
  Evaluation of the major complications (cardiopulmonary, stroke, wound complications)
Major complications | 1 month
  Major complications at 1 month
Hospital stay | Assessed at Discharge, approximately 3 days
  Total duration of hospital stay assessed at Discharge
Minor complications | 1 month
  Minor complications at 1 month
All cause mortality | 1 month
  All cause mortality at 1 month
Re operation | 1 month
  Re operation at 1 month
Re hospitalization | 1 month
  Re hospitalization at 1 month
Device related SAE | 1 month
  Device related SAE at 1 month
All AEs | 1 month
  All AEs at 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Robert Pflugmacher, Prof, Principal Investigator — University Hospital, Bonn
Locations (1):
- Universitätsklinikum Bonn, Bonn, Germany

REFERENCES:
- [Derived] Bornemann R, Himstedt J, Boszczyk B, Bowald S, Sander K, Mikulowski S, Farhoud HMES, Pflugmacher R. A Prospective Clinical Study to Evaluate Safety and Performance of an Intra-Surgical Hydraulic Distractor During Spinal Surgeries. Med Devices (Auckl). 2025 Oct 24;18:525-536. doi: 10.2147/MDER.S537601. eCollection 2025. PMID 41164796